CLINICAL TRIAL: NCT04475159
Title: Combined Neoadjuvant Systemic and PIPAC Therapy (NASPIT) for Patients With Colorectal Peritoneal Metastasis Eligible for CRS and HIPEC: A Prospective Phase II Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prof. Aviram Nissan (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Aviram Nissan, Proffesor, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6881-20-SMC
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Metastatic Colorectal Cancer; Peritoneal Carcinomatosis; Colon Adenocarcinoma
MeSH Terms: conditions — Colorectal Neoplasms; Peritoneal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PIPAC arm (Experimental): Together with neoadjuvant systemic therpay PIPAC will be performed twice and regional chemotherpay will be administered before planned CRS/HIPEC
  Interventions: Procedure: Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC)

INTERVENTIONS:
Procedure: Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) — Pressurized Intraperitoneal Aerosol Chemotherapy will be delivered to the abdominal cavity by means of laparoscopy.

SUMMARY:
Pressurized intraperitoneal aerosol chemotherapy (PIPAC) is a novel drug-delivery system developed to deliver, effectively and safely, small doses of cytotoxic agents into peritoneal tumor deposits. It is currently used for palliation and for down-staging of patients who are non-eligible for cytoreductive surgery (CRS) and hyperthermic intra-peritoneal chemotherapy (HIPEC).

The aim of this study is to evaluate the efficacy of PIPAC used in neoadjuvant setting to enhance the response of patients with colorectal peritoneal metastasis when combined with neoadjuvant systemic therapy for patients eligible to CRS/HIPEC prior to planned surgery.

DETAILED DESCRIPTION:
This is an open label, single arm, single center, phase II trial to study the added efficacy benefit of PIPAC administered in the neoadjuvant setting in combination with systemic therapy for patients eligible for CRS/HIPEC.

the following procedures will be done to all study population. Visit 0 (Week #0) screening - Clinical evaluation and baseline cross-sectional imaging. Patients will be evaluated for their eligibility and recruited if found suitable.

(Week #1) tumor board discussion to ensure eligibility and staging (Week #2-4) Initiation of systemic therapy, if not been already started (2 cycles): Systemic therapy will be administered and tailored by the treating oncologist as per patient tolerability. If already on chemotherapy at visit 0, patients will continue chemotherapy until first PIPAC.

Visit 1 (Week #4) first PIPAC: Diagnostic laparoscopy, staging, PCI evaluation and biopsies will be taken as described earlier.

Systemic therapy (2 cycles, Week #4-8): Systemic therapy will be administered and tailored by the treating oncologist as per patient tolerability.

Visit 2 (Week #6) - post first PIPAC - Surgical Oncology Clinic: evaluation of PIPAC tolerability and possible side effects or complications. Cross sectional imaging to monitor progression prior to the upcoming second PIPAC.

Visit 3 (Week #8) - second PIPAC: Diagnostic laparoscopy, staging, PCI evaluation and biopsies will be taken as described earlier.

Systemic therapy (2 cycles, Week #8-12): Systemic therapy will be administered and tailored by the treating oncologist as per patient tolerability. Systemic therapy will be stopped at week#12 (2-4 weeks) prior to planned CRS/HIPEC Visit 4 (Week #10) - post second PIPAC - Surgical Oncology Clinic: evaluation of PIPAC tolerability, quality of life, and possible side effects or complications after PIPAC.

Visit 5 (Week #12-14) - Surgical evaluation and cross-sectional imaging - Surgical Oncology Clinic: Planning for upcoming CRS/HIPEC Visit 6 (Week #14-16) - CRS/HIPEC: proper PCI evaluation, complete tumor cytoreduction and HIPEC will be targeted. The extent of surgery, technical difficulties including OR time and blood loss will be documented.

Visit 7 follow up visit: will be conducted within 1 month after hospital discharge. Tolerability and possible complications post-surgery will be evaluated.

Visit 8-11 follow up visits: Surgical Oncology Clinic evaluation: cross sectional imaging, Tumor markers and clinical evaluation will be conducted for any signs of possible recurrence on 3 monthly bases Visit 12-13 follow up: Surgical oncology clinic: cross sectional imaging, Tumor markers and clinical evaluation will be conducted for any signs of possible recurrence on 6 monthly bases. The follow up for the trial will be concluded at this stage (total of 3 years follow up).

To be noted that patient systemic chemotherapy would not be interrupted throughout the treatment protocol and PIPAC therapy will be delivered in-between chemotherapy cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study and must be willing to return for follow-up
3. 18 years of age or older.
4. Biopsy (histopathology or cytology) diagnosis of colorectal cancer as defined by the WHO or by cross-sectional imaging reviewed by a board-certified radiologist.
5. Good performance status (ECOG < 2), Karnofski >60.
6. Patients with low or acceptable surgical risk (American Society of Anesthesiology (ASA) score of 3 or less.
7. Patient is a candidate for CRS and HIPEC as discussed and recommended by the institutional disease management team (DMT, Tumor Board)
8. Patient receiving systemic chemotherapy for up to a maximum of 6 months from peritoneal diagnosis management with stable or responsive disease are eligible for the trial.
9. Absolute neutrophil count (ANC) exceeds 1200/mm3, white blood cell count exceeds 4000/mm3 and platelet count is greater than 100,000/mm3
10. An international normalized ratio (INR) ≤ 1.5 (patients who are therapeutically anticoagulated for non-related medical conditions such as atrial fibrillation and whose anti-thrombotic treatment can be withheld for operation will be eligible
11. Adequate hepatic function must be met as evidenced by total serum bilirubin ≤ 1.5 mg/dl (patients with total bilirubin > 1.5 mg/dL eligible only with Gilbert's syndrome); alkaline phosphatase < 2.5 times the upper limit of normal; and, AST less than 1.5 times upper limit of normal [alkaline phosphatase and AST cannot both exceed the upper limit of normal
12. Serum renal functional parameters, BUN and creatinine are within normal limits
13. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening or with negative pregnancy test at screening.
14. Life expectancy of at least six months

Exclusion Criteria:

1. Patients with unresectable (not eligible for CRS/HIPEC) tumors as decided by a multidisciplinary disease management team
2. Patients that already received multiple cycles of systemic chemotherapy of more than 6 months and or show progression of disease on systemic therapy.
3. Patients with extraperitoneal disease.
4. Pregnancy or lactation
5. Patients with low performance status (ECOG > 2 or Karnofski < 60%)
6. Any one or more of the following hematological abnormalities
7. Hgb < 8gm/dl unable to be corrected with transfusion
8. Absolute Neutrophil Count < 1200/mm3
9. White blood cell count < 4000/mm3
10. Platelet count < 100,000/mm3
11. INR > 1.5 (except in patients who are therapeutically AST anticoagulated for non-related medical conditions such as atrial fibrillation and whose anti-thrombotic treatment cannot be withheld for operation will be eligible)
12. History of hepatic cirrhosis or present hepatic dysfunction
13. Alkaline phosphatase ≥ 2.5 times the upper limit of normal
14. ≥ 1.5 times upper limit of normal
15. Serum bilirubin > 1.5 mg/dl (except for patients with Gilbert's syndrome who must have direct bilirubin ≤ 1.0 mg/dl)
16. Alkaline phosphatase and AST both exceed the upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Best Overall Response Rates (BORR) | 12 months after last patient recruitment
  Clinically, at time of laparoscopic exploration, tumor burden and distribution will be assessed. Peritoneal cancer index (PCI) will be documented. Final evaluation of tumor burden, PCI and clinical response will be evaluated at time of CRS/HIPEC. Radiologically, a baseline abdominal computed tomography (CT) scan will be acquired <4 weeks before the initiation of the treatment plan and will be repeated before CRS/HIPEC. Response will be evaluated by an independent radiologist as per RECIST criteria 1.1. Pathologically, biopsies from representative lesions will be taken. During the first procedure, before PIPAC delivery one sample from each abdominal quadrant and will be submitted to histopathology examination. Each biopsy site will be marked by a sliver clip for subsequent biopsies in the following PIPAC. Final pathological assessment will be done from specimens obtained at time of cytoreductive surgery .

SECONDARY OUTCOMES:
Recurrence free survival (RFS) | 3 years after the end of the trial
  Recurrence free survival (RFS) will be calculated from the date of CRS/HIPEC to the date of documented disease recurrence. Events for the RFS endpoint include clinical, radiological (CT, PET), serological (CEA, CA-19-9, CA-125) and/or surgical exploration.